CLINICAL TRIAL: NCT00333294
Title: A Phase II Open-Label Multicentre Study Of The Efficacy Of ZD1839 (IRESSA™) In Combination With Irradiation Followed By Chemotherapy In Patients With Inoperable Stage III Non Small Cell Lung Cancer
Brief Title: Phase II Iressa + Irradiation Followed by Chemo in NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0530
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Radiotherapy; Cisplatin; Vinorelbine

INTERVENTIONS:
Drug: Gefitinib
Procedure: Radiation therapy
Drug: Cisplatin
Drug: Vinorelbine

SUMMARY:
The objective of this study is to determine wether the ZD1839 associated with a radiotherapy, before the beginning of chemotherapy is effective in the treatment of your disease and to evaluate the tolerance of these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* 18 to 75 years inclusive.
* At least one measurable lesions histologically confirmed inoperable stage III NSCLC.
* WHO performance status of 0 to 2 inclusive.
* Adequate pulmonary function, pulmonary dose volume histogram less than or equal to 40 %.
* Life expectancy of at least 6 months.
* Using secure contraceptives precautions.

Exclusion Criteria:

* Any previous anti cancer therapy for NSCLC.
* Known severe hypersensitivity to these products
* Any evidence of clinically active interstitial lung disease
* Other co-existing malignancies, symptomatic metastases.
* Abnormal blood test
* Weight loss of over 15% in the 3 months before the start of the study.
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-09; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To estimate the objective response rate in patients treated with this drug

SECONDARY OUTCOMES:
Determine the safety and toxicity of this drug in these patients

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca France Medical Director, MD, Study Director — AstraZeneca
Locations (4):
- France (4):
  - Research Site, Clermont-Ferrand
  - Research Site, Grenoble
  - Research Site, Nantes
  - Research SIte, Paris